CLINICAL TRIAL: NCT03015844
Title: A Compassionate Use/Expanded Access Protocol Using 131I-MIBG Therapy for Patients With Refractory Neuroblastoma and Metastatic Pheochromocytoma
Status: Available | Type: Expanded Access
Sponsor: Northwell Health (Other)
Collaborators: Cohen Children's Medical Center (Other)
Responsible Party: Principal Investigator, Julie Krystal, Head, Early Phase Clinical Trials, Pediatric Hematology-Oncology, Northwell Health
Other Study IDs: CCMC1611
Record Dates: First submitted 2017-01-05; First posted 2017-01-10 (Estimated); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Neuroblastoma; Pheochromocytoma
Keywords: MIBG; 131I-MIBG; relapsed; neuroblastoma; pheochromocytoma
MeSH Terms: conditions — Neuroblastoma; Pheochromocytoma; Recurrence | interventions — 3-Iodobenzylguanidine

INTERVENTIONS:
Drug: 131-I-meta-iodobenzylguanidine
  Other Names: 131I-MIBG; Iobenguane

SUMMARY:
This is an expanded access protocol/compassionate use single institution study designed to determine the palliative benefit and toxicity of 131I-MIBG in patients with progressive neuroblastoma and metastatic pheochromocytoma who are not eligible for therapies of higher priority. Response rate, toxicity, and time to progression and death will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Relapsed/Refractory neuroblastoma, with an original diagnosis made histologically or from elevated urine catecholamines with abnormal tumor cells in bone marrow OR relapsed/refractory pheochromocytoma.
* Disease status: Progressive disease at any time (defined as any new lesion or an increase in size by >25% of pre-existing disease), or a failure to respond to standard therapy. Patients must have evidence of MIBG uptake into tumor at ≥ one site within 6 weeks prior to entry on study and subsequent to any intervening therapy
* Prior therapy: A minimum of two weeks since should have elapsed since any chemotherapy causing myelosuppression. It must be a minimum of three months since receiving radiation to any of the following fields: craniospinal, total abdominal, whole lung, total body irradiation. For any other sites of radiation, at least 2 weeks should have elapsed. For patients who received radiation to the only site of MIBG-avid disease within two months of study entry, biopsy confirmation of residual active disease is required, with positive bone marrow being sufficient. At least 7 days should have elapsed since completion of therapy with a biologic agent and at least 3 half-lives should have elapsed since therapy with a monoclonal antibody. No cytokine therapy may be given within 24 hours of receiving 131I-MIBG. Patients may have received prior MIBG therapy, provided they demonstrated a response or stable disease initially, with progressive disease occurring at least 35 days following treatment.
* Organ function: ANC >500/uL, platelets >20,000/uL with transfusion allowed. Bilirubin ≤2x ULN, AST/ALT ≤10x ULN.Serum Creatinine ≤2x ULN OR 24-hour creatinine clearance OR GFR ≥60ml/min/1.73m2. Normal lung function demonstrated by no dyspnea, exercise intolerance or oxygen requirement. Oxygen saturation ≥94% on room air. No clinically significant cardiac dysfunction and ejection fraction ≥45% on echocardiogram.
* Stem cells: Patients must have a minimum of 2.0 x106/kg viable CD34+ peripheral blood stem cells for re-infusion following 131I-MIBG. An additional back-up of 2.0x106/kg CD34+ cells is recommended but not required.
* Life expectancy longer than 8 weeks,Karnofsky or Lansky performance status of ≥ 50%

Exclusion Criteria:

* Pregnant or lactating patients
* Disease of any organ system that would compromise the patient's ability to participate in the study, including hemodialysis. Significant organ impairment should be discussed with the Principal Investigator prior to study entry
* Patients with active grade 3-4 infection, as defined by the NCI CTCAE V4.0.
* Patients with known MBIG-avid brain parenchymal disease (leptomeningeal or skull based metastases are eligible).
* In patients with metastatic pheochromocytoma, a urinalysis must be preformed prior to study enrollment. If proteinuria is present, a 24 hour urine must be collected and total protein determined. If the 24-hour urine protein is above the institutional upper limit of normal, the patient is excluded.

Ages: 365 Days to 29 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Cohen Children's Medical Center, New Hyde Park, New York, United States

REFERENCES:
- [Background] Matthay KK, Quach A, Huberty J, Franc BL, Hawkins RA, Jackson H, Groshen S, Shusterman S, Yanik G, Veatch J, Brophy P, Villablanca JG, Maris JM. Iodine-131--metaiodobenzylguanidine double infusion with autologous stem-cell rescue for neuroblastoma: a new approaches to neuroblastoma therapy phase I study. J Clin Oncol. 2009 Mar 1;27(7):1020-5. doi: 10.1200/JCO.2007.15.7628. Epub 2009 Jan 26. PMID 19171714
- [Background] Kang TI, Brophy P, Hickeson M, Heyman S, Evans AE, Charron M, Maris JM. Targeted radiotherapy with submyeloablative doses of 131I-MIBG is effective for disease palliation in highly refractory neuroblastoma. J Pediatr Hematol Oncol. 2003 Oct;25(10):769-73. doi: 10.1097/00043426-200310000-00005. PMID 14528098
- [Background] Yanik GA, Levine JE, Matthay KK, Sisson JC, Shulkin BL, Shapiro B, Hubers D, Spalding S, Braun T, Ferrara JL, Hutchinson RJ. Pilot study of iodine-131-metaiodobenzylguanidine in combination with myeloablative chemotherapy and autologous stem-cell support for the treatment of neuroblastoma. J Clin Oncol. 2002 Apr 15;20(8):2142-9. doi: 10.1200/JCO.2002.08.124. PMID 11956276
- [Background] Matthay KK, DeSantes K, Hasegawa B, Huberty J, Hattner RS, Ablin A, Reynolds CP, Seeger RC, Weinberg VK, Price D. Phase I dose escalation of 131I-metaiodobenzylguanidine with autologous bone marrow support in refractory neuroblastoma. J Clin Oncol. 1998 Jan;16(1):229-36. doi: 10.1200/JCO.1998.16.1.229. PMID 9440747
- [Background] Matthay KK, Yanik G, Messina J, Quach A, Huberty J, Cheng SC, Veatch J, Goldsby R, Brophy P, Kersun LS, Hawkins RA, Maris JM. Phase II study on the effect of disease sites, age, and prior therapy on response to iodine-131-metaiodobenzylguanidine therapy in refractory neuroblastoma. J Clin Oncol. 2007 Mar 20;25(9):1054-60. doi: 10.1200/JCO.2006.09.3484. PMID 17369569